CLINICAL TRIAL: NCT04570228
Title: Clinical Evaluation of the Therapeutic Intra-Vascular Ultrasound (TIVUS™) System for Pulmonary Artery Denervation in Patients With Pulmonary Arterial Hypertension
Brief Title: TROPHY PAH Pivotal Study - TReatment of Pulmonary HYpertension for PAH Pivotal Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SoniVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLNS03-001 - TROPHY 3 Protocol
Record Dates: First submitted 2020-09-08; First posted 2020-09-30 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:1 with a sham controlled arm, with subjects and all follow up staff blinded to the subject treatment. Subjects will be unblinded at 6M, and sham control group will be offered treatment at this time if they meet the inclusion/ exclusion criteria. The primary effectiveness endpoint is measured at 6 months. The safety endpoint for blinded patients is at 6 months, and for treated patients again at 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment group (Active Comparator): Pulmonary artery denervation with the TIVUS™ System will be performed immediately after the right heart catheterization and pulmonary artery angiography.
  Interventions: Device: Pulmonary artery denervation
- Sham control group (Sham Comparator): A sham treatment of pulmonary artery denervation with the TIVUS™ System will be performed immediately after the right heart catheterization pulmonary artery angiography. The sham procedure will be identical to the denervation procedure, with the only exception that the procedure will use a sham setting on the control console.
  Interventions: Device: Sham procedure

INTERVENTIONS:
Device: Pulmonary artery denervation — The TIVUS system will be used for pulmonary artery denervation using non focused ultrasound
  Arms: Treatment group
Device: Sham procedure — A sham procedure would be performed using the TIVUS system without delivering the non focused ultrasound
  Arms: Sham control group

SUMMARY:
Theis is a prospective, multicenter, blinded, randomized sham controlled pivotal clinical trial with a crossover at 6M, to assess the safety and effectiveness of pulmonary artery denervation with the TIVUS™ System in subjects with PAH. The study will assess improved and/or maintained exercise tolerance in patients with PAH through the analysis of exercise tolerance, hemodynamic changes, clinical worsening and the quality of life who got treated by the TIVUS system.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent to participate in the study obtained from the subject, according to local regulations, prior to initiation of any study mandated procedure.
2. Male or female ≥ 18 years of age at the time of screening
3. Subject with known pulmonary arterial hypertension (PAH), which has been diagnosed as idiopathic PAH, connective tissue disease PAH, anorexigen induced, familial PAH or corrected congenital heart defects more than 1 year prior to enrollment, confirmed by right heart catheterization performed prior to screening and showing all of the following:

   * Mean pulmonary artery pressure (mPAP) ≥25 mmHg at rest
   * Pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤15 mmHg
   * Pulmonary vascular resistance (PVR) at rest >3 Wood units (240 dyne*s/cm^5)
4. Subject is on maximally tolerated medical therapy for PAH, as determined by his PAH physician
5. Subject is adhering to a stable drug regimen (i.e., with no changes of dose or medication for a minimum of 3 months prior to enrollment)
6. Subject is able to tolerate IV contrast used for the angiograms during treatment
7. Subject is WHO functional class II or III

Exclusion Criteria:

1. Subject is treated with parenteral prostanoids and has not been on a stable dose for at least 3 months
2. Subjects with portal-pulmonary hypertension, Group 2, 3 and 4 PH
3. Pregnant women or women planning a pregnancy within 12 months of study enrolment
4. Subject with significant co-morbid conditions which, at the discretion of the PI, are deemed to prohibit study entry
5. Subject with life expectancy of less than a year
6. Concurrent enrollment in another device or drug trial except for observational studies (unless specifically approved by the sponsor)
7. Subject with pulmonary artery anatomy that precludes treatment with the TIVUS System
8. Subject who has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident in the previous 6 months
9. Subject experiencing a current episode of acute decompensated heart failure
10. Subject who has cardiac pacemakers/ICD/CRT-D that were implanted fewer than three months prior to enrollment.
11. Subject who has implantable Cardiomems device, or other implanted device that might be contraindicated for therapeutic ultrasound energy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
6 minute walking distance (6MWD) | 6 months
  Statistical difference in 6MWD between the treated group and the sham control group
The rate of procedure and treatment related SAEs reported | 12 months

SECONDARY OUTCOMES:
Statistical difference between the treated group and the sham control group in exercise tolerance as measured using the change in activity parameters using the Actigraph Centrepoint watch | 6 months
Difference between time to clinical worsening event between the treated group and the sham control group | 6 months
Difference between the number of clinical worsening events between the treated group and the sham control group | 6 months
  The definition of clinical worsening events includes: all cause death, hospitalization for worsening PAH, lung/heart transplant, arterial septostomy, initiation of parenteral prostanoid therapy, change in dose and/or number of PAH specific medication. Each event will be counted as a single event and per each patient the total number of events will be recorded
Difference between the treated group and the sham control group in resting mean right atrial pressure (mRAP) | 6 months
Difference between the treated group and the sham control group in resting mean pulmonary artery pressure (mPAP) | 6 months
Difference between the treated group and the sham control group in resting pulmonary vascular resistance (PVR) | 6 months
Difference between the treated group and the sham control group in resting cardiac index (CI) | 6 months
Difference between the treated group and the sham control group in Quality of Life (QOL) score using the SF36 questionnaire | 6 months
  The SF36 is a 0-100 score, the lower the score is the lower the quality of life is, so that zero is equivalent to maximum disability and a score of 100 is equivalent to no disability at all
Difference between the treated group and the sham control group of NT-pro-BNP levels | 6 months
Difference between the treated group and the sham control group in patients' clinical pulmonary arterial hypertension condition defined by worsening of World Health Organization (WHO) functional class | 6 months
  PAH patient's WHO functional class is a scale of 1 to 4 based on the symptoms patient experience when doing everyday activities, were Functional Class 1 and 2 are associated with limited effect on patient activity and lower risk status, and Functional Class 3 and 4 are associated with limited activity and higher risk status
Percent of patients who improve or maintain their exercise tolerance (as measured by 6MWD and actigraphy) | 6 months

OTHER OUTCOMES:
Clinical change of pulmonary arterial hypertension condition defined by escalation of PAH specific drug therapy | 6, 12, 24, 36 month
  Change in the dose of medication
Clinical change of pulmonary arterial hypertension condition defined by escalation of PAH specific drug therapy | 6, 12, 24, 36 month
  Change in the number of PAH specific medication
Clinical change of pulmonary arterial hypertension condition defined by escalation of concomitant drug therapy | 6, 12, 24, 36 month
  Change in the number of concomitant medication
Clinical change of pulmonary arterial hypertension condition defined by escalation of concomitant drug therapy | 6, 12, 24, 36 month
  Change in dose of a medication
Clinical change of pulmonary arterial hypertension condition defined by change from baseline of ECG parameters demonstrating initiation or worsening of heart block | 6, 12, 24, 36 month
  Heart block is defined as long PR interval, wide or narrow QRS complex and/or QRS complex in various leads are oriented rightward and anteriorly. Heart block will be noted as either present or not present. Any change from baseline will be noted.
Clinical change of pulmonary arterial hypertension condition defined by change from baseline of ECG parameters indicating initiation or worsening of arrhythmia | 6, 12, 24, 36 month
  Arrhythmia is defined when the P-P interval and/or R-R interval has differences of more than 10% and/or there are no visible P waves and/or irregularly irregular QRS complex is present. Arrhythmia will be noted as either present or not present. Any change from baseline will be noted.
Clinical change of pulmonary arterial hypertension condition defined by change from baseline of ECG parameters indicating initiation or worsening of right ventricular hypertrophy (RVH) | 6, 12, 24, 36 month
  Right ventricular hypertrophy is when the following are present: right axis deviation > 90 degrees, tall R-waves in RV leads; deep S-waves in LV leads, slight increase in QRS duration and ST-T changes directed opposite to QRS direction (i.e., wide QRS/T angle). Right ventricular hypertrophy will be noted as either present or not present. Any change from baseline will be noted.
Clinical change of pulmonary arterial hypertension condition defined by change from baseline of ECG parameters indicating initiation or worsening of axis deviation | 6, 12, 24, 36 month
  Axis deviation is present when QRS axis is greater than +90° or smaller than +30°. Axis deviation will be noted as either present or not present. Any change from baseline will be noted.
Change from baseline of 6MWD | 12, 24, 36 month
Change from baseline of NT-pro BNP levels | 12, 24, 36 month
Change from baseline of actigraphy measures as will be measured using an Actigraph Centrepoint Insight Activity monitor | 12, 24, 36 month
Change from baseline of Quality of Life (QOL) score using the SF36 questionnaire | 12, 24, 36 month
  PAH patient's WHO functional class is a scale of 1 to 4 based on the symptoms patient experience when doing everyday activities, were Functional Class 1 and 2 are associated with limited effect on patient activity and lower risk status, and Functional Class 3 and 4 are associated with limited activity and higher risk status
Survival or the cause of mortality | 6, 12, 24, 36 month
Amount of Hospitalizations events due to pulmonary arterial hypertension | 6, 12, 24, 36 month
Number of patients with clinical worsening of PAH condition resulting with interventional or surgical procedures, such as heart/lung transplant or atrial septostomy. | 6, 12, 24, 36 month
Clinical change of pulmonary arterial hypertension condition defined by worsening of patients' WHO functional class | 12, 24, 36 month
  PAH patient's WHO functional class is a scale of 1 to 4 based on the symptoms patient experience when doing everyday activities, were Functional Class 1 and 2 are associated with limited effect on patient activity and lower risk status, and Functional Class 3 and 4 are associated with limited activity and higher risk status
Clinical change of pulmonary arterial hypertension condition defined by escalation of concomitant drug therapy | 6, 12, 24, 36 month
  Change in the dose of medication
Clinical change of pulmonary arterial hypertension condition defined by escalation of concomitant drug therapy | 6, 12, 24, 36 month
  Change in the number of concomitant medications